CLINICAL TRIAL: NCT00096746
Title: An Exploratory Study of the Effect of the Atazanavir (ATV) I50L Mutation on Subsequent Treatment Response
Brief Title: Effect of the Atazanavir (ATV) 150L Mutation on Subsequent Treatment Response in HIV Infected Subjects
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Other Study IDs: AI424-079
Record Dates: First submitted 2004-11-15; First posted 2004-11-16 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infection
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A1: HIV infected individuals on first line ATV based HAART with presence of I50L mutation.
  Interventions: Drug: LPV/RTV + 2NRTIs
- A2: HIV infected PI naïve on failed NNRTI based regimen.
  Interventions: Drug: LPV/RTV + 2NRTIs

INTERVENTIONS:
Drug: LPV/RTV + 2NRTIs — Tablets, Oral, Variable, Twice daily, 48 weeks.
  Groups: A1
Drug: LPV/RTV + 2NRTIs — Tablets, Oral, Variable, Twice daily, 48 weeks.
  Groups: A2

SUMMARY:
This study will compare the response of subjects who failed a first-line ATV-containing regimen and who have the 150L-containing virus to subsequent protease inhibitor (PI)-containing therapy with that of a cohort who has failed a first-line reverse transcriptase inhibitor (NNRTI), and is subsequently receiving PI-containing therapy.

ELIGIBILITY:
Inclusion Criteria:

* Currently on a first-line antiretroviral regimen containing ATV with a confirmed rebound and a genotype that verifies the presence of an 150L mutation OR on a first-line regimen containing an NNRTI and PI-naive, with a confirmed rebound

Exclusion Criteria:

* Women of child bearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 8 weeks after the study.
* Women who are pregnant or breastfeeding.
* A life expectancy of <12 months.
* Presence of a newly diagnosed HIV-related opportunistic infection or any other medical condition requiring acute therapy at the time of enrollment.
* Active alcohol or substance abuse sufficient, in the investigator's opinion, to prevent adequate adherence to study therapy or to increase the risk of developing pancreatitis or chemical hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected individuals on first line ATV based HAART with presence of I50L mutation & HIV infected PI naïve on failed NNRTI based regimen.
Sampling Method: Non-Probability Sample
Enrollment: 200
Dates: Start 2004-11; Primary Completion 2006-09 (Actual); Study Completion 2006-09

PRIMARY OUTCOMES:
The log10 HIV RNA change from baseline for each cohort. | through Week 48

SECONDARY OUTCOMES:
Evaluate proportion of patients with plasma HIV RNA <50 copies/mL | at Weeks 24, 48, 72, and 96.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Chair — Bristol-Myers Squibb
Locations (37):
- United States (13):
  - Local Institution, Phoenix, Arizona
  - Local Institution, Altamonte Springs, Florida
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Vero Beach, Florida
  - Local Institution, Honolulu, Hawaii
  - Local Instution, Wichita, Kansas
  - Local Instution, Lexington, Kentucky
  - Local Institution, Louisville, Kentucky
  - Local Institution, East Orange, New Jersey
  - Local Institution, Albany, New York
  - Local Institution, Huntersville, North Carolina
  - Local Institution, Portland, Oregon
  - Local Institution, Dallas, Texas
- Argentina (7):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, La Plata, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, Buenos Aires
- Brazil (5):
  - Local Institution, Curitiba, Paraná
  - Local Institution, Recife, Pernambuco
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Campinas, São Paulo
  - Local Institution, São Paulo
- Local Institution, Guatemala City, Guatemala
- Mexico (2):
  - Local Institution, Durango, Durango
  - Local Institution, Guadalajara, Jalisco
- Local Institution, Lima, Lima Province, Peru
- South Africa (8):
  - Local Institution, Port Elizabeth, Eastern Cape
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Bedford Gardens, Gauteng
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Meadowdale, Gauteng
  - Local Institution, Westdene, Gauteng
  - Local Institution, Mowbray, Western Cape
  - Local Institution, Rugby, Western Cape